CLINICAL TRIAL: NCT01741662
Title: Prevalence of Psychocognitive Impairments in Adolescents Surviving Childhood Leukemia : LEA-PsyCog
Acronym: LEA-PsyCog
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2012-A01129-34; 2012-29 (Other: AP HM)
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Adolescents Surviving Childhood Leukemia LEA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- group psychopathological (Other)
  Interventions: Other: neuropsychological evaluation

INTERVENTIONS:
Other: neuropsychological evaluation

SUMMARY:
The objective of the LEA-PsyCog project is to assess the prevalence of psychiatric disorders and psychocognitive impairments in adolescents surviving childhood leukemia .

The second objective is to explore the complex relationships between psycocognitive development and soiciodemodemographics data, main characteristics of leukemia, treatments, side-effects, quality of life and characteristics of proxyies environment.

3. Materials and Methods The LEA study is based on the constitution of a multi-centric prospective cohort in 11 university hospitals: Bordeaux, Clermont-Ferrand, Grenoble, Lyon, Paris (Trousseau, Robert Debré, St Louis), Marseille, Montpellier, Nancy, Nice, Rennes. Are inclued in LEA all the children diagnosed and treated for acute leukemia since January 1980 (incident and prevalent cases), surviving at month 24 for the AML and ALL grafted in complete remission and at month 48 for the ALL not grafted in first complete remission.

The LEA Psy-Cog study rests on a sample of the LEA cohort. Are included the patients 12-17-years-old from the PACA-Corse sub-cohort (administrative district of 4 million of people which corresponds to the Marseille and Nice centers). Patients from this two centers are the patients with the more important length of survey, allowing us to produce a not biaised estimation of prevalence rate. Finally, the choice of this subsample is supported by the proximity of the Mediterranean Center for Adolescent in Marseilles, specifically dedicated to the psychological follow-up of children suffering from cancer.

ELIGIBILITY:
Inclusion Criteria:

* - Age 18-year-old subordinate at the time of the diagnosis;
* Diagnosis of acute(sharp) leukaemia;
* Diagnosis from January, 1980;
* Treatment(Processing) of the acute(sharp) leukaemia introduced in one of the inquiring centers (services(departments) specialized hematology and Clermont Ferrand's pediatric oncology, Grenoble, Lyon, Marseille, Nancy, Nancy, Nice, Paris - Robert Debré/Saint Debré/Saint Louis/Trousseau Louis/Trousseau;
* Living in France;
* Possessing a national insurance scheme
* 24-month-old Survivor of recoil(drop) with regard to(compared with) the diagnosis for the Leukaemia Aiguës Myéloblastiques (LAM) and Leukaemia Aiguës Lymphoblastiques ( LAL) transplanted in 1st complete forgiveness; or in 48 months of recoil(drop) with regard to(compared with) the diagnosis for the LAL not transplanted in first complete forgiveness;

Exclusion Criteria:

* Failure to respect the criteria of inclusion beforehand quoted,
* Initial Treatment(Processing) realized except 2 participating centers (Marseille, Nice), even in case of moving in in the geographical zones covered by these centers during the phase of treatment(processing) or in the course of follow-up

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 170 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Diagnosis psychopathological | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France